CLINICAL TRIAL: NCT01592812
Title: Investigation of the Arterial Effects of the Veinoplus(r) Stimlator Device.
Brief Title: Arterial Inflow and Muscle Ischemia During Calf Stimulation With the Veinoplus Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A01546-35
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electrical stimulation (Experimental): Evaluation of the effect of calf stimulation on flow and tissue oxygenation
  Interventions: Device: electrical muscle stimulation

INTERVENTIONS:
Device: electrical muscle stimulation — Duration of the stimulation 20 minutes
  Other Names: Veinoplus device

SUMMARY:
Stimulation of arterial inflow to the lower limb is important to obtain functional improvement in peripheral artery diseased (PAD) patients with claudication. The clinical effect of muscle stimulation to increase arterial inflow and the direct evaluation of the regional blood flow impairment (RBFI) in the area of stimulation, have not been evaluated in PAD patients.

Fifteen adult patients with stable arterial claudication will participate. Recruitment will be performed among patients referred for exercise oxymetry (treadmill: 3.2km.h-1, 10% slope) After two minutes of rest, the gastrocnemius will be stimulated for 20 minutes at an increasing frequency rate with 5 min steps (1 Hz, 1.25 Hz, 1.5 Hz and 1.75 Hz) on the most symptomatic side.

The investigators record the tcpo2 value, arterial blood inflow with ultrasound of the femoral artery, and near infra-red spectrometry (NIRS) on both sides.

Patients will be instructed to report eventual contraction-induced pain in the stimulated calf.

DETAILED DESCRIPTION:
Investigations are conducted in an air-conditioned 22+/-2 °C room, with the patient comfortably seated on an armchair.

Measured ware started at rest and performed throughout the period pf stimulation and for 10 minutes after the end of the stimulation

Muscle stimulation:

We apply a series of 20 minutes of stimulation with the Veinoplus® device. The device delivers a stimulation of incremental rate with 5 minutes intervals, with 1 Hz, 1.25 Hz, 1.5 Hz and 1.75 Hz and then stops automatically.

Ultrasound measurements The Diameter of the superficial femoral artery was measured at rest on both sides before each study. The VTI of 3 cardiac cycles (three peaks systolic velocity) will be measured by duplex ultrasound imaging, to calculate the arterial inflow to the leg. Results will be expressed in l /min.

Tcpo2 recording TcpO2 is measured at the chest and on both calves with TCM 400 (Radiometer, DK). Results are expressed in DROP index(mmHg) values.

Near Infra-red spectroscopy (NIRS) We use the ARTinis NIRS device (ARTinis; NL) to estimate tissue saturation (StO2) on both gastrocnemius muscles of the leg.

Systemic hemodynamic parameters

Systemic and diastolic arterial pressures and heart rate are recorded every two minutes using Dinamap V100 (GE france).

ELIGIBILITY:
Inclusion Criteria:

* French native
* Stable stage 2 peripheral artery disease
* Patent femoral artery on both sides
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* Adults protected by maw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
arterial inflow | during stimulation
  Ultrasound and doppler measurement of femoral inflow before, during and for 10 minutes after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, MD; PhD, Principal Investigator — University Hospital in Angers (France)
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Abraham P, Mateus V, Bieuzen F, Ouedraogo N, Cisse F, Leftheriotis G. Calf muscle stimulation with the Veinoplus device results in a significant increase in lower limb inflow without generating limb ischemia or pain in patients with peripheral artery disease. J Vasc Surg. 2013 Mar;57(3):714-9. doi: 10.1016/j.jvs.2012.08.117. Epub 2013 Jan 9. PMID 23312939